CLINICAL TRIAL: NCT03402412
Title: Atopic Dermatitis: Early Gene Expression Changes as Predictors of Therapeutic Response to Narrow-band UVB Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jan Øivind Holm, Associate Professor and Consultant Dermatologist, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/466
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Arm (Experimental): Narrow-band UVB will be given to a small part of the patients skin with eczema. The rest of the skin surface serves as control.
  Interventions: Other: narrow-band UVB

INTERVENTIONS:
Other: narrow-band UVB — Standard established treatment for atopic dermatitis with narrow-band UVB will be used in this study but initially only on a small amount of skin to assess what changes takes place in the skin.

SUMMARY:
Phototherapy with narrow band (nb) ultraviolet B (UVB) is a safe and effective but time consuming treatment option for patients with widespread eczema. Despite efficacy we know little about how it works, and even less why some patients fail to respond. Tintle et al showed that nb-UVB induced strong suppression of the Th2 and Th22 axes in patients with atopic dermatitis (AD), and also normalized the epidermal barrier function. We want to map the very early changes in gene expression after UVB-treatment in order to shed light on disease mechanisms, which eventually could lead to better treatment options.

DETAILED DESCRIPTION:
Patients will be scored with Patient-Oriented Eczema Measure (POEM), Eczema Area and Severity Index (EASI), SCORAD (SCORing Atopic Dermatitis) and Dermatology Life Quality Index (DLQI) to assess disease severity. The investigators will measure trans epidermal water loss (TEWL), take bacterial swabs for analysis of the microbiome and culture for Staphylococcus aureus and test for mutations in the filaggrin-gene by sputum samples. Blood serum samples will be taken to measure serum (s) -Immunoglobulin E, s-vitamin D status, full blood count including white cell differential and different cytokines. Any history of allergic asthma, allergic rhinitis or food allergy will be noted as well as any recent history of sun exposure, use of tanning beds or UVB-therapy.

The suberythemal dose of UVB for each patient will be established. In each patient two contralateral areas (e.g. both underarms) with eczema will be chosen, which are as similar as possible regarding distribution and severity. One area will be biopsied with a 4mm punch followed by locally treatment with nb-UVB (311nm) three times. In this way the untreated side will serve as an internal control. Both sides will be biopsied after these initial three rounds of treatment. The patients will then undergo 24 standard full-body nb-UV-treatment sessions followed by a new biopsy of the same area. Skin from non-lesional sun-protected skin from nates will also be samples prior to and after UVB-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis

Exclusion Criteria:

* Other inflammatory skin disease
* Concurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Early gene expression changes in atopic skin after UVB-treatment | Study period for each participant: 9 weeks
  Gene expression changes

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Oivind Holm, MD, PhD, Principal Investigator — Oslo University Hospital/University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tintle S, Shemer A, Suarez-Farinas M, Fujita H, Gilleaudeau P, Sullivan-Whalen M, Johnson-Huang L, Chiricozzi A, Cardinale I, Duan S, Bowcock A, Krueger JG, Guttman-Yassky E. Reversal of atopic dermatitis with narrow-band UVB phototherapy and biomarkers for therapeutic response. J Allergy Clin Immunol. 2011 Sep;128(3):583-93.e1-4. doi: 10.1016/j.jaci.2011.05.042. Epub 2011 Jul 16. PMID 21762976